CLINICAL TRIAL: NCT01385592
Title: 12-week, Double-blind, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of AFQ056 in Reducing Moderate to Severe L-dopa Induced Dyskinesias in Patients With Parkinson's Disease
Brief Title: Evaluation of the Efficacy and Safety of AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2222; 2011-002073-30 (EudraCT Number)
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-03

CONDITIONS: Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders
Keywords: Parkinson Disease; L-dopa; Levodopa; Dyskinesia; Anti-Dyskinesia Agents
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Movement Disorders; Parkinsonian Disorders | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AFQ056 100 mg (Experimental)
  Interventions: Drug: AFQ056
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056
  Arms: AFQ056 100 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of AFQ056 in patients that have Parkinson's Disease L-dopa Induced Dyskinesias (PD-LID)

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with Parkinson's disease (PD), treated with L-Dopa, experiencing dyskinesias for at least three months
* Outpatients who are on a stable anti-parkinsonian treatment regimen for at least four weeks

Exclusion Criteria:

* Surgical treatment for PD
* Cancer within the past 5 years (other than localized skin cancer and prostate cancer that has been effectively treated)
* Advanced, severe or unstable disease (other than PD) or evidence of dementia that may interfere with the study outcome evaluations

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Anti-dyskinetic efficacy as measured by the modified AIMS (Abnormal Involuntary Movement Scale) total score. To assess how titration of AFQ056 at 2-week intervals affects tolerability profile | 12 weeks

SECONDARY OUTCOMES:
Anti-dyskinetic efficacy as measured by the Lang-Fahn Activities of Daily Living Dyskinesia Scale (LFADLDS) | 12 weeks
Change from baseline on patient's disability caused by the dyskinesia as assessed by a clinician-rated global impression of change (CGIC) | 12 weeks
Total ON- and OFF-times and ON-time with dyskinesia and with troublesome dyskinesias (patient diary) | 12 weeks
Anti-dyskinetic efficacy as measured by items 32, 33 and 34 of Part IV of the Unified Parkinson's Disease Rating Scale (UPDRS ) | 12 weeks
Safety of AFQ056 as measured by changes in vital signs, laboratory values, electrocardiogram and number of Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (2):
  - Novartis Investigative Site, Sunnyvale, California
  - Novartis Investigative Site, Englewood, Colorado
- Canada (2):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
- France (4):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
- Germany (9):
  - Novartis Investigative Site, Beelitz-Heilstätten
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Westerstede/Oldenburg
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
- Italy (3):
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Spain (4):
  - Novartis Investigative Site, Sant Cugat del Vallès, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Madrid

REFERENCES:
- [Derived] Trenkwalder C, Stocchi F, Poewe W, Dronamraju N, Kenney C, Shah A, von Raison F, Graf A. Mavoglurant in Parkinson's patients with l-Dopa-induced dyskinesias: Two randomized phase 2 studies. Mov Disord. 2016 Jul;31(7):1054-8. doi: 10.1002/mds.26585. Epub 2016 May 23. PMID 27214258
- See also: Results for CAFQ056A2222 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9863